CLINICAL TRIAL: NCT05076201
Title: Process of Regulation in Addictions: Vulnerability Emotional Factors to Craving
Acronym: Procrav
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Ramsay santé (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-A01248-49
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Craving; Emotional Dysfunction; Self-Regulation, Emotion; Alexithymia; Cocaine Addict
Keywords: vulnerability
MeSH Terms: conditions — Emotional Regulation; Affective Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with completed rehab (Experimental): The aim of this research is to follow-up a cohort of patients at the end of their detoxification cure (cocaïne).
  Interventions: Behavioral: Patients with completed rehab

INTERVENTIONS:
Behavioral: Patients with completed rehab — The main objective is to measure the level of cocaine craving, 6 months after the end of their detoxification treatment (outpatient or full hospitalization), in patients with a diagnosis of moderate to severe dependence (DSM 5) to cocaine and co-addiction, or not, to alcohol and / or psychostimulants. To evaluate cocaïne craving,the questionnaire CCQ-Brief will be used.

SUMMARY:
The aim of this study is to have a better understanding of the relationship between self-controle difficulties (and more specifically the inhibition deficit in impulsivity), emotional regulation disorders such as alexithymia and craving.This study will be the first in France to specify the interactions between self-regulkation processes dysfunctions and emotional dysfunctions in craving.

DETAILED DESCRIPTION:
The main objective is to measure the level of cocaine craving, 6 months after the end of their detoxification treatment (outpatient or full hospitalization), in patients with a diagnosis of moderate to severe dependence (DSM 5) to cocaine and co-addiction, or not, to alcohol and / or psychostimulants. To evaluate cocaïne craving,the questionnaire CCQ-Brief will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patient, men or women between 18 and 60 years-old
* Patient with a diagnosis of moderate to severe dependence (DSM 5) to cocaine with or without co-addictions to alcohol or psychostimulant.
* Patient on day-hospitalisation or full hospitalisation
* Patient affiliated or beneficiary to a social security scheme.
* Patient having signed the free and informed consent.

Exclusion Criteria:

* Patient with psychiatric disorders psychosis type
* Patient with severe chronic somatic disease.
* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, breastfeeding or parturient woman.
* Patient hospitalized without consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Cocaïne craving evaluation | 6 months
  Using the French version of the questionnaire CCQ-Brief "Cocaïne Craving Questionnaire".

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique privée, Marseille, France